CLINICAL TRIAL: NCT07015541
Title: Effects of Quadriceps Focused Interventions in Adolescent With ACL Reconstruction
Brief Title: Quadriceps Strengthening ACL Reconstruction
Acronym: ACL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexandra Abbott, Clinical Assistant Professor (Orthopedic Surgery), Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 80260
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional neuromuscular electrical stimulation (NMES) and blood flow restriction (BFR) (Experimental): Participants receive a 6-week NMES intervention from week 1 to week 6 post-surgery, followed by a 10-week BFR intervention from week 7 to week 16. Participants also receive standard rehabilitation care as part of their routine postsurgical recovery process.
  Interventions: Other: NMES and BFR; Other: Standard physical therapy
- Standard rehabilitation (Active Comparator): Participants receive standard rehabilitation care as part of their routine postsurgical recovery process.
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Other: NMES and BFR — NMES is applied when patients perform quadriceps strengthening exercises. BFR is applied during compound exercises.
  Arms: Additional neuromuscular electrical stimulation (NMES) and blood flow restriction (BFR)
Other: Standard physical therapy — Standard physical therapy (week 1-16) includes interventions for typical impairments following ACLR. The initial phase will focus on pain and effusion control, restoration of knee range of motion, followed by gait normalization, lower extremity strength training, then running and plyometrics.

SUMMARY:
The purpose of this study is to investigate the effects of quadriceps focused interventions on knee function and biomechanics in adolescent patients with anterior cruciate ligament reconstruction (ACLR)

ELIGIBILITY:
Inclusion Criteria:

* no history of knee injury/surgery of the contralateral limb

Exclusion Criteria:

* (1) bilateral knee injuries
* (2) prior knee ligament injury and/or surgery
* (3) multiple ligament injuries and/or ruptures
* (4) conditions in which NMES and BFR are contraindicated

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Peak force as measured by isometric knee extension force test | 16 weeks post surgery
  Isometric knee extension force will be measured with a dynamometer.
Force steadiness as measured by isometric knee extension force test | 16 weeks post surgery
  Isometric knee extension force will be measured with a dynamometer

SECONDARY OUTCOMES:
Sagittal plane peak angle at the hip during countermovement jump landing | 16 weeks post surgery
  Motion analysis will be conducted using the cloud-based OpenCap application
Sagittal plane peak angle at the knee during countermovement jump landing | 16 weeks post surgery
  Motion analysis will be conducted using the cloud-based OpenCap application
Sagittal plane peak angle at the ankle during countermovement jump landing | 16 weeks post surgery
  Motion analysis will be conducted using the cloud-based OpenCap application

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M Abbott, MD, Principal Investigator — Stanford School of Medicine
Locations (1):
- Stanford Medicine Children's Health, Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohta H, Kurosawa H, Ikeda H, Iwase Y, Satou N, Nakamura S. Low-load resistance muscular training with moderate restriction of blood flow after anterior cruciate ligament reconstruction. Acta Orthop Scand. 2003 Feb;74(1):62-8. doi: 10.1080/00016470310013680. PMID 12635796
- [Background] Kim KM, Croy T, Hertel J, Saliba S. Effects of neuromuscular electrical stimulation after anterior cruciate ligament reconstruction on quadriceps strength, function, and patient-oriented outcomes: a systematic review. J Orthop Sports Phys Ther. 2010 Jul;40(7):383-91. doi: 10.2519/jospt.2010.3184. PMID 20592480